CLINICAL TRIAL: NCT03247881
Title: Pilot Study on Mixed Nuts and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS57
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nut Free Diet (Other): Participants will consume whatever they like, as much as they like, from a pre-determined buffet with 0 g/d of mixed nuts.
  Interventions: Other: Nut Free Diet
- Added Mixed Nuts Diet (Active Comparator): Participants will consume whatever they like, as much as they like, from a pre-determined buffet which will include 2 servings (2 ounces) of mixed nuts per day (1 serving just prior to breakfast and 1 serving as an afternoon snack).
  Interventions: Other: Added Mixed Nuts Diet

INTERVENTIONS:
Other: Nut Free Diet — Participants will consume whatever they like, as much as they like, from a pre-determined buffet with 0 g/d of mixed nuts.
  Other Names: Control Diet
  Arms: Nut Free Diet
Other: Added Mixed Nuts Diet — Participants will consume whatever they like, as much as they like, from a pre-determined buffet which will include 2 servings (2 ounces) of mixed nuts per day (1 serving just prior to breakfast and 1 serving as an afternoon snack).
  Arms: Added Mixed Nuts Diet

SUMMARY:
The objectives of this study are 1) to determine if consumption of mixed nuts influences food intake and choice, and 2) to determine how personality traits affect food choice, including mood, stress, tendency to seek approval, tendency toward food cravings, and approach to food intake control.

DETAILED DESCRIPTION:
The condition of being overweight or obese has skyrocketed in recent decades, bringing with it many secondary health problems. Therefore, it is important to seek strategies to promote weight loss and to assist in weight maintenance after weight loss. Different diet compositions may have different effects on satiety and thus affect food choice. A pilot study will be conducted to determine if mixed nuts affect food selection and intake. Questionnaires will also be administered to determine if personality characteristics are also influencing food choice.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 60 Years Old
* 5 year cancer-free

Exclusion Criteria:

* pregnant, lactating, or intending to become pregnant during the study
* known allergy to study foods, including nuts
* use of tobacco products
* history of bariatric surgery or nutrient malabsorption disease or diseases requiring special diet
* Crohn's disease or diverticulitis
* suspected or known strictures, fistulas, or physiological/mechanical GI obstruction
* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Self report of alcohol or substance abuse within the past 12 months and/or current acute treatment or participation in a rehabilitation program for those problems (long-term participation in Alcoholics Anonymous is not an exclusion)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Body Mass will be measured | Day 0, prior to beginning the diet, day 8, day 29, and day 60
  To track the change in body mass, subjects will be weighed on a scale.

SECONDARY OUTCOMES:
Questionnaires will be administered | Once during the study, no specific time.
  Questionnaires addressing control of eating, eating attitude, social approval, and social desirability will be administered.
Mood questionnaire will be administered | Day 0, Day 8, and Day 29.
  A mood questionnaire will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, Principal Investigator — USDA-ARS, Beltsville Human Nutrition Research Center
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No